CLINICAL TRIAL: NCT03679884
Title: Multi-center, Double-blind, Parallel-group, Randomized, Placebo-controlled, Three Doses, 40-week Extension to Studies ID-078A301 and ID-078A302 to Assess the Long Term Safety and Tolerability of ACT-541468 in Adult and Elderly Subjects With Insomnia Disorder
Brief Title: Study to Assess the Long Term Safety and Tolerability of ACT-541468 (Daridorexant) in Adult and Elderly Subjects Suffering From Difficulties to Sleep
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-078A303
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — daridorexant

STUDY DESIGN:
Intervention Model Description: Multi-center, double-blind, parallel-group, randomized, placebo-controlled, three doses, 40-week extension study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Daridorexant 10 mg (Experimental): Film-coated tablets administered orally, once daily in the evening
  Interventions: Drug: Daridorexant 10 mg
- Daridorexant 25 mg (Experimental): Film-coated tablets administered orally, once daily in the evening
  Interventions: Drug: Daridorexant 25 mg
- Daridorexant 50 mg (Experimental): Film-coated tablets administered orally, once daily in the evening
  Interventions: Drug: Daridorexant 50 mg
- Placebo (Placebo Comparator): Film-coated tablets administered orally, once daily in the evening
  Interventions: Drug: Placebo
- Ex-Placebo Daridorexant 25 mg (Experimental): Film-coated tablets administered orally, once daily in the evening
  Interventions: Drug: Daridorexant 25 mg

INTERVENTIONS:
Drug: Daridorexant 10 mg — Daridorexant 10 mg film-coated tablets
  Arms: Daridorexant 10 mg
Drug: Daridorexant 25 mg — Daridorexant 25 mg film-coated tablets
  Arms: Daridorexant 25 mg; Ex-Placebo Daridorexant 25 mg
Drug: Daridorexant 50 mg — Daridorexant 50 mg film-coated tablets
  Arms: Daridorexant 50 mg
Drug: Placebo — Matching placebo film-coated tablets
  Arms: Placebo

SUMMARY:
Study to assess the long term safety and tolerability of daridorexant in adult and elderly subjects suffering from difficulties to sleep

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure (Visit 1).
* Having completed the DB study treatment and the run-out period of ID-078A301 (NCT03545191) or ID-078A302 (NCT03575104).
* For woman of childbearing potential, the following is required:

  * Negative urine pregnancy test (EOT of ID-078A301 or ID-078A302 studies)
  * Agreement to use the contraception scheme as required by the protocol from Visit 1 up to at least 30 days after EODBT.

Exclusion Criteria:

* Unstable medical condition, significant medical disorder or acute illness, C-SSRS©, ECG, hematology or biochemistry test results in ID-078A301 and ID-078A302, which in the opinion of the investigator could affect the subject's safety or interfere with the study assessments (Visit 1).
* For female subjects: lactating or planning to become pregnant during the duration of the study (Visit 1).
* Positive urine drug test (for benzodiazepines, barbiturates, cannabinoids, opiates, amphetamines, or cocaine) or presence of alcohol in exhaled breath as detected by breathalyzer test (EOT of ID-078A301 or ID-078A302 studies if same day as Visit 1 or Visit 1 if within 7 days after EOT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (106):
- United States (53):
  - Pulmonary Associates of the Southeast/WCR, Birmingham, Alabama
  - Pulmonary Associates, Pa, Glendale, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Preferred Research Partners, Inc, Little Rock, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Core Healthcare Group, Cerritos, California
  - Marvel Clinical Research, Huntington Beach, California
  - Clinical Trials Research, Lincoln, California
  - Long Beach Clinical Trials, Long Beach, California
  - Artemis Institute For Clinical Research - Riverside, Riverside, California
  - Artemis institute for Clinical Research, San Diego, California
  - Pacific Research Network, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Santa Monica Clinical Trials, Santa Monica, California
  - Empire Clinical Research, Upland, California
  - Innovative Clinical Research, Lafayette, Colorado
  - PAB Clinical Research, Brandon, Florida
  - St. Francis Sleep Allergy and Lung Institute, Clearwater, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Research Centers of America, Hollywood, Florida
  - Canvas Clinical Research, LLC, Lake Worth, Florida
  - BioMed Research Institute, Miami, Florida
  - Clinical Research Group of St. Petersburgh, St. Petersburg, Florida
  - Clinical Site Partners, LLC, Winter Park, Florida
  - Neurotrials Research Incorporated, Atlanta, Georgia
  - Sleep Practitioners, LLC, Macon, Georgia
  - Saltzer Clinical Research, Nampa, Idaho
  - Helene Emsellem, MD, Chevy Chase, Maryland
  - Sleep Disorders Center of the Mid-Atlantic, Glen Burnie, Maryland
  - Infinity Medical Research, Inc., North Dartmouth, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - Barrett Clinic, La Vista, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Clinilabs NYC, New York, New York
  - Research Carolina of Hickory, Hickory, North Carolina
  - Research Carolina of Huntersville, Huntersville, North Carolina
  - Coastal Carolina Healthcare, New Bern, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Clinical Trials of America - NC, LLC, Winston-Salem, North Carolina
  - CTI Clinical Research II, Cincinnati, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Aventiv Research Inc., Dublin, Ohio
  - Cleveland Sleep Research Center, Middleburg Heights, Ohio
  - Oregon Center for Clinical Investigations,Inc, Salem, Oregon
  - Brian Abaluck LLC, Paoli, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - FutureSearch Trials of Neurology, LP, Austin, Texas
  - Inquest Clinical Research, Baytown, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Jacksonville Center for Clinical Research, Jacksonville, Texas
  - Sleep Disorders Centers of the Mid-Atlantic, Vienna, Virginia
  - Swedish Medical Center, Seattle, Washington
- Hospital UZ Leuven_ Pneumology Department, Leuven, Belgium
- Acibadem City Clinic Tokuda Hospital EAD, Sofia, Bulgaria
- Canada (7):
  - Queensway Sleep Lab Sleep Clinic (MedSleep), Etobicoke
  - The Medical Arts Health Research Group, Kelowna
  - Somni Research Inc., Markham
  - CRIUSMQ- CIUSSSCN, CETS (clinique du sommeil), Québec
  - CANADIAN PHASE ONWARD INC. (Toronto), Toronto
  - MedSleep, Toronto
  - Jodha Tishon Inc., Toronto
- Scan Sleep Specialists, Copenhagen, Denmark
- Finland (4):
  - Vitalmed Uniklinikka, Helsinki
  - Oivauni Oy - Kuopio, Kuopio
  - Oivauni Oy - Tampere, Tampere
  - Unitutkimusyksikkö, Turun Yliopisto, Turku
- CHU NIMES - Unité de Sommeil, Nîmes, France
- Germany (22):
  - St Hedwig-Krankenhaus, Klinik für Schlaf- und Chronomedizin, Berlin
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - emovis GmbH, Berlin
  - Charité - Universitätsmedizin Berlin - Campus Benjamin Franklin Kompetenzzentrum Schlafmedizin, Berlin
  - Synexus Berlin Research Centre, Berlin
  - Synexus Clinical Research GmbH, Bochum
  - Klinische Forschung Dresden GmbH, Dresden
  - Klinik imd Poliklinik fur Neurochirurgie, Dresden
  - Synexus Clinical Research GmbH, Frankfurt
  - Clinical Trial Center North GmbH & Co. KG, Hamburg
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Klinische Forschung Hannover Mitte GmbH, Hanover
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe
  - Studienzentrum Wilhelmshöhe GmbH, Kassel
  - Synexus Leipzig Research Centre, Leipzig
  - Zentrum für Integrative Psychiatrie (ZiP) Universität zu Lübeck, Lübeck
  - Central Insitute of Mental Health Sleep laboratory Medical Faculty Mannheim/Heidelberg University, Mannheim
  - Klinikum Rechts der lsar TU München Dept. of Psychiatry and Psychotherapy, München
  - Klinik und Poliklinik für Psychiatrie, Psychosomatik und Psychotherapie der Universität am Bezirksklinikum Regensburg, Regensburg
  - SOMNIBENE Institut für Medizinische Forschung und Schlafmedizin Schwerin GmbH, Schwerin
  - Kinische Forschung Schwerin GmbH, Schwerin
  - ZMS Zentrum für medizinische Studien GmbH, Warendorf
- Hungary (2):
  - Magyar Honvédség Egészségügyi Központ, Neurológiai Osztály, Budapest
  - Somnius Kft. SomnoCenter Szeged, Szeged
- Poland (3):
  - PI-House - Centrum Badań Klinicznych, Gdansk
  - Ośrodek Medycyny Study Nurseu Instytutu Psychiatrii i Neurologii (Sleep Disorders Center), Warsaw
  - EMC Instytut Medyczny SA, Przychodnia przy Łowieckiej, Wroclaw
- South Korea (2):
  - 4F Neuroimaging analysis laboratory, 56 Dalseong-ro, Jung-gu, Daegu
  - 2F Psychiatry Outpatient, 93, Jungbu-daero, Paldal-gu, Suwon
- Spain (5):
  - Centro Médico Teknon - Medicina del Sueño, Barcelona
  - Hospital Universitari Vall d'Hebron - Neurophisiology Deparment - Sleep Unit, Barcelona
  - Instituto de Investigaciones del Sueno, Madrid
  - Hospital Universitario Araba - Unidad Funcional de Trastornos del Sueño, Vitoria-Gasteiz
  - Hospital MAZ - Neurophisiology and Sleep Department, Zaragoza
- Sweden (3):
  - Göteborgs Universitet, Centrum för sömn och vakenhetsstörningar, Gothenburg
  - Universitetssjukhuset Örebro Neurokliniken, Sömnenheten, Örebro
  - Sömnutredningsmottagningen, smärtcentrum Akademiska sjukhuset, Uppsala
- Zentrum für Schlafmedizin Zürcher Oberland, Zürcher RehaZentrum Wald, Wald, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dutta S, Singhal S, Shah R, Charan J, Dhingra S, Haque M. Daridorexant as a novel pharmacotherapeutic approach in insomnia: a systematic review and meta-analysis. Expert Opin Drug Saf. 2023 Jul-Dec;22(12):1237-1251. doi: 10.1080/14740338.2023.2243217. Epub 2023 Aug 7. PMID 37526060
- [Derived] Kunz D, Dauvilliers Y, Benes H, Garcia-Borreguero D, Plazzi G, Seboek Kinter D, Coloma P, Rausch M, Sassi-Sayadi M, Thein S. Long-Term Safety and Tolerability of Daridorexant in Patients with Insomnia Disorder. CNS Drugs. 2023 Jan;37(1):93-106. doi: 10.1007/s40263-022-00980-8. Epub 2022 Dec 9. PMID 36484969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety-four sites in 14 countries (Belgium, Bulgaria, Canada, Denmark, Finland, France, Germany, Hungary, South Korea, Poland, Spain, Sweden, Switzerland, and the US) enrolled and randomized subjects.
Pre-assignment Details: Subjects assigned to the daridorexant arms in Study ID-078A301 and 302 received the same dose in the ID-078A303 extension study. Subjects assigned to the placebo arm in Study ID-078A301 and 302 were re-randomized to receive either placebo or 25 mg daridorexant in a 1:1 ratio, with treatment allocation stratified by age into 2 categories (< 65 and ≥ 65 years).
  Note: Subjects' demographic and baseline characteristics were collected in the respective confirmatory 12-week study (ID-078A301 or 302).
Groups:
- Daridorexant 10 mg: Film-coated tablets administered orally, once daily in the evening
  Daridorexant 10 mg: Daridorexant 10 mg tablets
- Daridorexant 25 mg; ExPlacebo/Daridorexant 25 mg: Film-coated tablets administered orally, once daily in the evening
  Daridorexant 25 mg: Daridorexant 25 mg tablets
- Daridorexant 50 mg: Film-coated tablets administered orally, once daily in the evening
  Daridorexant 50 mg: Daridorexant 50 mg tablets
- Placebo: Film-coated tablets administered orally, once daily in the evening
  Placebo: Daridorexant matching placebo tablets
Period: Overall Study
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Daridorexant 50 mg | Placebo | ExPlacebo/Daridorexant 25 mg
Started (DB treatment period) | 142 | 268 | 137 | 128 | 126
Completed (DB treatment period) | 99 | 190 | 93 | 78 | 90
Not Completed | 43 | 78 | 44 | 50 | 36
Not completed — Other | 12 | 12 | 12 | 7 | 8
Not completed — Lack of Efficacy | 15 | 29 | 13 | 29 | 10
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 10 | 9 | 6 | 6
Not completed — Withdrawal by Subject | 12 | 23 | 8 | 8 | 9
Not completed — Lost to Follow-up | 1 | 4 | 2 | 0 | 3

BASELINE CHARACTERISTICS:
Population: These are the participants included in the FAS. The discrepancy with previous table (Participant Flow) is due to 3 subjects on FAS (2 on daridorexant 25 mg and 1 on ex-placebo/ daridorexant 25 mg) not starting DB treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Daridorexant 50 mg | Placebo | ExPlacebo/Daridorexant 25 mg | Total
Number analyzed (Participants) | 142 | 270 | 137 | 128 | 127 | 804
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 80 | 166 | 83 | 70 | 70 | 469
  >=65 years | 62 | 104 | 54 | 58 | 57 | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (12.8) | 57.6 (14.1) | 56.9 (13.6) | 59.2 (12.6) | 56.5 (15.5) | 57.7 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 199 | 98 | 92 | 83 | 575
  Male | 39 | 71 | 39 | 36 | 44 | 229
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Black or African American | 6 | 19 | 15 | 8 | 7 | 55
    American Indian or Alaska Native | 2 | 0 | 1 | 0 | 0 | 3
    Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
    Asian | 5 | 8 | 0 | 2 | 5 | 20
    White | 128 | 243 | 121 | 115 | 115 | 722
    Other | 0 | 0 | 0 | 2 | 0 | 2
    Not permitted as per legislation/regulation | 1 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 6 | 33 | 19 | 10 | 13 | 81
    Not Hispanic or Latino | 135 | 237 | 118 | 118 | 114 | 722
    Unknown | 0 | 0 | 0 | 0 | 0 | 0
    Not permitted as per legislation/regulation | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Total no. of Subjects With at Least One TEAE
Description: The primary objective of the study was to assess the long-term safety and tolerability of 10, 25 and 50 mg daridorexant.
  The total no. of subjects with at least one TEAE is presented here; no statistical analysis was conducted.
  The full set of safety data is available in the Section "Adverse events".
Time Frame: TEAEs (AEs that started or worsened during the double-blind study period up to 30 days after double-blind study treatment end date) are reported. Total duration: up to 44 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- ExPlacebo / Daridorexant 25 mg: Film-coated tablets administered orally, once daily in the evening
  Daridorexant 25 mg: Daridorexant 25 mg tablets
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Daridorexant 50 mg | Placebo | ExPlacebo / Daridorexant 25 mg
Number analyzed (Participants) | 142 | 268 | 137 | 128 | 126
Participants | 53 | 103 | 55 | 45 | 48

ADVERSE EVENTS:
Time Frame: All treatment-emergent SAEs and AEs are reported.
Description: TEAEs (AEs that started or worsened during the double-blind study period up to 30 days after double-blind study treatment end date) are reported. Total duration: up to 44 weeks.
Groups:
- Ex-Placebo Daridorexant 25 mg: Film-coated tablets administered orally, once daily in the evening
  Daridorexant 25 mg: Daridorexant 25 mg tablets
Arm/Group | Daridorexant 10 mg | Daridorexant 25 mg | Daridorexant 50 mg | Placebo | Ex-Placebo Daridorexant 25 mg
All-Cause Mortality (participants affected / at risk) | 1/142 | 1/268 | 0/137 | 0/128 | 0/126
Serious Adverse Events (participants affected / at risk) | 5/142 | 12/268 | 7/137 | 2/128 | 4/126
Other Adverse Events (participants affected / at risk) | 7/142 | 15/268 | 12/137 | 6/128 | 11/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daridorexant 10 mg (N=142) | Daridorexant 25 mg (N=268) | Daridorexant 50 mg (N=137) | Placebo (N=128) | Ex-Placebo Daridorexant 25 mg (N=126)
Aortic valve disease mixed (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis subacute (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daridorexant 10 mg (N=142) | Daridorexant 25 mg (N=268) | Daridorexant 50 mg (N=137) | Placebo (N=128) | Ex-Placebo Daridorexant 25 mg (N=126)
Nasopharyngitis (Infections and infestations) | 7 (10) | 15 (16) | 12 (13) | 6 (6) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Idorsia for review at least 30 days prior to submission for publication or presentation at a congress. Upon review, Idorsia may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights. Neither the institution nor the investigator should permit publication during such a review period.

DOCUMENTS (3):
  • Study Protocol: Study Protocol (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT03679884/Prot_000.pdf
  • Study Protocol: Study Protocol Addendum (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT03679884/Prot_001.pdf
  • Statistical Analysis Plan (2020-06-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT03679884/SAP_002.pdf